CLINICAL TRIAL: NCT05865054
Title: A Longitudinal Study of Orbital and Cranial Vessel Wall MRI in Giant Cell Arteritis by the Vascular MRI Evaluation in Giant Cell Arteritis (VEGA) Collaborative
Brief Title: Vascular MRI Evaluation in Giant Cell Arteritis (VEGA)
Acronym: VEGA
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Rennie Rhee, M.D., MSCE, Assistant Professor of Medicine, University of Pennsylvania
Other Study IDs: 843171; R01AR084199-01A1 (NIH)
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Giant Cell Arteritis
Keywords: Temporal Arteritis; Horton's Giant Cell Arteritis; Horton's Disease; Horton Giant Cell Arteritis; Horton Disease; Cranial Arteritis
MeSH Terms: conditions — Giant Cell Arteritis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Ocular GCA: GCA with clinical diagnosis of ischemic optic neuropathy or other ocular condition
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI)
- Non-Ocular GCA: GCA without ocular manifestations
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI)
- Non-GCA: Initially suspected to have GCA but final clinical diagnosis not GCA
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) — Combined orbital and cranial vessel wall MRI

SUMMARY:
The research study is being conducted to determine the utility of magnetic resonance imaging (MRI) in identifying inflammation of arteries supplying blood to the head, brain, and eyes. The target population includes patient with suspected giant cell arteritis (GCA; temporal arteritis).

DETAILED DESCRIPTION:
After signing the consent form, participants will complete an MRI scan within 2 weeks of enrollment and fill out questionnaires related to their disease. Follow up visits and MRI scans may occur at 6-months after the initial MRI scan or at the time of relapse.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or older
* First presentation of suspected GCA
* New or worsening cranial manifestations within 4 weeks of enrollment concerning for active GCA
* Elevated CRP greater than 1.0 mg/dl
* Plan to undergo temporal artery biopsy or ultrasound for diagnosis

Exclusion Criteria:

* Contra-indication to receiving MRI including:

Implanted medical devices, pacemaker, and metallic foreign fragments inside body/orbits Known gadolinium allergy Women who are pregnant or nursing

* Absence of cranial symptoms related to GCA (e.g., only large vessel GCA)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the ambulatory clinic, emergency department, or inpatient settings.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2033-07 (Estimated)

PRIMARY OUTCOMES:
Vessel Wall Enhancement Score | Up to 12 months
  Enhancement of cranial vessel wall, orbital structures, or other cranial structures. Scores range from 0 to 3; 0 being no inflammation and 3 being more enhancement or inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Rennie Rhee, MD, Principal Investigator — University of Pennsylvania
Locations (4):
- United States (2):
  - Mayo Building and Gonda Building, Rochester, Minnesota
  - 3400 Civic Center Blvd, Philadelphia, Pennsylvania
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada
- University Hospital Wuerzburg, Würzburg, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: No
This has not been approved by the ethics committee at some sites.